CLINICAL TRIAL: NCT02680769
Title: Daily Supplementation of Magnesium Citrate in Moderate-severe Chronic Obstructive Pulmonary Disease: a Randomized, Controlled, Double-blind Trial
Brief Title: Effect of Magnesium Supplementation in COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3577
Record Dates: First submitted 2016-02-08; First posted 2016-02-12 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium (Experimental): 300 mg of citrate Mg/daily
  Interventions: Dietary Supplement: 300 mg of citrate Mg
- Placebo (Placebo Comparator): placebo group
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: 300 mg of citrate Mg — This group will take an oral supplementation of 300 mg of citrate magnesium
  Arms: Magnesium
Other: Placebo — This group will take a placebo
  Arms: Placebo

SUMMARY:
Magnesium (Mg) is involved in several pathways that could be affected in chronic obstructive pulmonary diseases (COPDs), namely in the contractility and excitability of neuro-muscolar endothelial cells and low-grade inflammation, a typical state of COPD. In this sense, several randomized controlled trials (RCTs) confirmed a positive role of Mg in asthma since long-period oral supplementation of Mg leads to a clinical and spirometric improvement.

Subjects with COPD seem to have a reduced bioavailability of Mg probably due to the use of drugs that may increase Mg losses (e.g. beta-agonists and cortisones), to a reduced dietary Mg intake, and heavy smoking. A recent study showed that the administration of endovenous or aerosol Mg sulphate with beta-agonists acutely improve maximum expiratory flow during COPD relapses as well as the prolonged treatment with endovenous sulphate Mg led to a reduction in pulmonary hyperinflation and increase in muscles involved in respiration, with a consequent clinical and instrumental improvement.

These evidences suggest that a chronic supplementation with Mg could improve COPD in clinical and instrumental parameters, but, at the best of our knowledge, no study was available in this sense.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years).
* Moderate-severe COPD (FEV1 between 30-80% of theorical values).

Exclusion Criteria:

* Already taking magnesium or calcium supplementations.
* Severe renal (creatinine clearance< 30 ml/min) or hepatic decline or presence of other co-morbidities interfering with outcomes (e.g. dementia).
* Hypermagnesemia (serum Mg>1.85 mmol/L).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Change in forced expiratory volume in the 1st second between baseline and 6 months | 0-3-6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Padova-Geriatrics Section, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gontijo-Amaral C, Ribeiro MA, Gontijo LS, Condino-Neto A, Ribeiro JD. Oral magnesium supplementation in asthmatic children: a double-blind randomized placebo-controlled trial. Eur J Clin Nutr. 2007 Jan;61(1):54-60. doi: 10.1038/sj.ejcn.1602475. Epub 2006 Jun 21. PMID 16788707
- [Result] Beasley R, Aldington S. Magnesium in the treatment of asthma. Curr Opin Allergy Clin Immunol. 2007 Feb;7(1):107-10. doi: 10.1097/ACI.0b013e328012ce4b. PMID 17218820
- [Result] Aziz HS, Blamoun AI, Shubair MK, Ismail MM, DeBari VA, Khan MA. Serum magnesium levels and acute exacerbation of chronic obstructive pulmonary disease: a retrospective study. Ann Clin Lab Sci. 2005 Autumn;35(4):423-7. PMID 16254259
- [Derived] Zanforlini BM, Ceolin C, Trevisan C, Alessi A, Seccia DM, Noale M, Maggi S, Guarnieri G, Vianello A, Sergi G. Clinical trial on the effects of oral magnesium supplementation in stable-phase COPD patients. Aging Clin Exp Res. 2022 Jan;34(1):167-174. doi: 10.1007/s40520-021-01921-z. Epub 2021 Jul 14. PMID 34260036